CLINICAL TRIAL: NCT02504372
Title: A Randomized, Phase 3 Trial With Anti-PD-1 Monoclonal Antibody Pembrolizumab (MK-3475) Versus Placebo for Patients With Early Stage NSCLC After Resection and Completion of Standard Adjuvant Therapy (PEARLS)
Brief Title: Study of Pembrolizumab (MK-3475) vs Placebo for Participants With Non-small Cell Lung Cancer After Resection With or Without Standard Adjuvant Therapy (MK-3475-091/KEYNOTE-091)
Acronym: PEARLS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ETOP (Unknown); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-091; EORTC-1416-LCG (Other: EORTC); 163457 (Registry Identifier: JAPIC-CTI); MK-3475-091 (Other: MSD); KEYNOTE-091 (Other: MSD); 2023-509137-39-00 (Registry Identifier: EU CT); U1111-1309-6051 (Registry Identifier: UTN); 2015-000575-27 (EudraCT Number)
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Results first posted 2024-02-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer (NSCLC); Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand (PDL)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg, intravenously (IV), every 3 weeks, for one year (expected maximum 18 doses).
  Interventions: Biological: Pembrolizumab
- Placebo (Placebo Comparator): Participants receive placebo, IV, every 3 weeks, for one year (expected maximum 18 doses).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab
Other: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
In this study, participants with Stage IB/II-IIIA non-small cell lung cancer (NSCLC) who have undergone surgical resection (lobectomy or pneumonectomy) with or without adjuvant chemotherapy will be treated with pembrolizumab or placebo. The primary study hypothesis is that pembrolizumab will provide improved disease-free survival (DFS) versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of NSCLC confirmed at surgery, any histology. Participants with two synchronous primary non-small cell lung cancers are excluded from the study
* Union for International Cancer Control (UICC) v7 Stage IB with T ≥ 4 cm, II-IIIA NSCLC after complete surgical resection with resection margins proved microscopically free of disease (R0). Carcinoma in situ can be present at the bronchial margin
* Available tumor sample obtained at surgical resection for programmed cell death ligand-1 (PD-L1) Immunohistochemistry (IHC) expression assessment
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Adequate organ function performed within 10 days of treatment initiation
* Female participants of childbearing potential must have a negative urine or serum pregnancy test at screening (within 72 hours of first infusion of study medication). If the urine test cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the participant to be eligible
* Female participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity starting with the first infusion of study treatment through 120 days after the last infusion of study treatment
* Female participants who are breast feeding must discontinue nursing prior to the first infusion of study medication and until 120 days after the last infusion study treatment
* Male participants must agree to use an adequate method of contraception starting with the first infusion of study treatment through 120 days after the last infusion of study treatment
* Absence of severe comorbidities that in the opinion of the Investigator might hamper the participation to the study and/or the treatment administration
* No prior or planned neo-adjuvant or adjuvant radiotherapy and/or neo-adjuvant chemotherapy for the current malignancy is allowed

Exclusion Criteria:

* Evidence of disease at clinical examination and/or baseline radiological assessment as documented by contrast enhanced chest/upper abdomen CT scan, brain CT/MRI and clinical examination
* More than 4 cycles of adjuvant therapy
* Prior treatment with anti-programmed cell death (anti-PD)-1, anti-PD ligand-1/2, anti-CD137, or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) modulators or any other immune-modulating agents
* Live vaccine within 30 days prior to the first infusion of study treatment
* Current participation or treatment with an investigational agent or use of an investigational device within 4 weeks of the first infusion of study treatment
* History of Human Immunodeficiency Virus (HIV) (known HIV 1/2 antibodies positive). No known active Hepatitis B or C
* Chronic use of immunosuppressive agents and/or systemic corticosteroids or any use in the last 3 days prior to the first infusion of study treatment
* History of interstitial lung disease or (non-infectious) pneumonitis that required oral or IV steroids (other than COPD exacerbation) or current pneumonitis
* Active autoimmune disease that has required systemic treatment in past 2 years
* History of a hematologic or primary solid tumor malignancy, unless in remission for at least 5 years with the exception of pT1-2 prostatic cancer Gleason score < 6, superficial bladder cancer, non melanomatous skin cancer or carcinoma in situ of the cervix
* Previous allogeneic tissue/solid organ transplant
* Active infection requiring therapy
* Surgery- or chemotherapy-related toxicity (non-hematological) not resolved to Grade 1 with the exception of alopecia, fatigue, neuropathy and lack of appetite /nausea
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last infusion of study treatment
* Participant will not be eligible if the participant is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or Sponsor staff directly involved with this trial, unless prospective site Review Board approval is given allowing exception to this criterion for a specific participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2026-01-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] O'Brien M, Paz-Ares L, Marreaud S, Dafni U, Oselin K, Havel L, Esteban E, Isla D, Martinez-Marti A, Faehling M, Tsuboi M, Lee JS, Nakagawa K, Yang J, Samkari A, Keller SM, Mauer M, Jha N, Stahel R, Besse B, Peters S; EORTC-1416-LCG/ETOP 8-15 - PEARLS/KEYNOTE-091 Investigators. Pembrolizumab versus placebo as adjuvant therapy for completely resected stage IB-IIIA non-small-cell lung cancer (PEARLS/KEYNOTE-091): an interim analysis of a randomised, triple-blind, phase 3 trial. Lancet Oncol. 2022 Oct;23(10):1274-1286. doi: 10.1016/S1470-2045(22)00518-6. Epub 2022 Sep 12. PMID 36108662
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant randomized to the study in error did not provide informed consent and was not included. No data was collected on this participant.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg, intravenously (IV), every 3 weeks, for one year.
- Placebo: Participants received placebo, IV, every 3 weeks, for one year.
Period: Overall Study
Arm/Group | Pembrolizumab | Placebo
Started | 590 | 587
Treated | 580 | 581
Completed | 0 | 0
Not Completed | 590 | 587
Not completed — Death | 136 | 154
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal of consent | 25 | 16
Not completed — Participants ongoing | 429 | 415

BASELINE CHARACTERISTICS:
Population: All randomized participants. One participant randomized to the study in error did not provide informed consent and was not included. No data was collected on this participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Placebo | Total
Number analyzed (Participants) | 590 | 587 | 1177
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.5) | 64.5 (8.4) | 64.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 184 | 373
  Male | 401 | 403 | 804
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 107 | 107 | 214
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 450 | 455 | 905
  More than one race | 10 | 3 | 13
  Unknown or Not Reported | 22 | 19 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease Stage at Baseline [Count of Participants; unit: Participants] — Participants were classified per American Joint Committee on Cancer Manual Edition 7th (AJCC V7) based on TNM classification where T refers to size and extent of primary tumor and if it invaded nearby tissue, N refers to location of nearby lymph nodes that have cancer and M refers to distant metastasis (spread of cancer to other parts). In stages I, II and III the cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues. In stage IV, the cancer has spread to distant parts of the body. Higher numbers mean the cancer is more advanced.
  Participants
    Stage IB | 85 | 87 | 172
    Stage II | 330 | 338 | 668
    Stage IIIA | 175 | 160 | 335
    Stage IV | 0 | 2 | 2
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Expression Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression status by immunohistochemistry assay using tumor tissue from a biopsy. Participants with a tumor proportion score (TPS) were classified as follows: <1% = PD-L1 negative, 1-49% = PD-L1 weakly positive; and ≥50% = PD-L1 strongly positive.
  Participants
    TPS <1% | 233 | 232 | 465
    TPS 1-49% | 189 | 190 | 379
    TPS ≥50% | 168 | 165 | 333
Adjuvant Chemotherapy at Baseline [Count of Participants; unit: Participants] — Participants were classified per receiving of standard adjuvant chemotherapy at baseline: Yes or No.
  Participants
    Yes | 506 | 504 | 1010
    No | 84 | 83 | 167
Geographic region [Count of Participants; unit: Participants] — Participants were classified based on their geographic region as those from: Western Europe, Easter Europe, Asia and Rest of the world.
  Participants
    Western Europe | 303 | 301 | 604
    Eastern Europe | 116 | 113 | 229
    Rest of the World | 65 | 68 | 133
    Asia | 106 | 105 | 211
Tumor Histology [Count of Participants; unit: Participants] — Participants were classified according to tumor histology: Squamous or Non-squamous. The tumor histology determined potential treatment regimen.
  Participants
    Squamous | 192 | 224 | 416
    Non-squamous | 398 | 363 | 761
Smoking status [Count of Participants; unit: Participants] — Participants were classified per centers of disease control and prevention (CDC) as: Never smoker (smoked fewer than 100 cigarettes in his/her lifetime), former smoker (smoked at least 100 cigarettes in his or her lifetime but who had quit smoking at the time of interview. and current smoker (smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes) at baseline.
  Participants
    Never smoker | 87 | 66 | 153
    Former smoker | 428 | 431 | 859
    Current smoker | 75 | 90 | 165

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS)
Description: DFS was defined as the time from randomization to either the date of disease recurrence or death (whatever the cause) as assessed by the investigator. Recurrence of disease was defined as local regional recurrence, a distant (metastatic) recurrence, or a second primary cancer. Occurrence of a second extra-pulmonary malignancy was considered to be an event.
Time Frame: Up to approximately 84 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 590 | 587
Months | 53.8 [46.2 to 67.0] | 43.0 [35.0 to 51.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.68 to 0.96] — HR and 95% confidence interval (95%CI) were based on multivariate Cox regression model with treatment adjusted by stage, PD-L1 status, adjuvant chemotherapy, region, histology, and smoking status

2. Primary Outcome: DFS in Programmed Death Ligand-1 (PDL-1) Strong Positive Participants With Tumor Proportion Score (TPS) ≥50%
Description: DFS in PDL-1 strong positive participants with TPS ≥50% was defined as the time from randomization to either the date of disease recurrence or death (whatever the cause) as assessed by the investigator. Recurrence of disease was defined as local regional recurrence, a distant (metastatic) recurrence, or a second primary cancer. Occurrence of a second extra-pulmonary malignancy was considered to be an event.
Time Frame: Up to approximately 84 months
Population: All randomized PDL-1 strong positive participants with TPS ≥50%. One participant randomized to the study in error did not provide informed consent and was not included. No data was collected on this participant.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 168 | 165
Months | 67.0 [47.8 to NA] — NA = Upper limit DFS was not reached at the time of last disease assessment due to insufficient number of participants with events. | 47.6 [36.4 to NA] — NA = Upper limit DFS was not reached at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Other; p = 0.13499, Regression, Cox; One-sided p-value was based on the permutation test with multivariate Cox regression model; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.59 to 1.16] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: DFS in PDL-1 Strong Positive Participants With TPS ≥1%
Description: DFS in PDL-1 strong positive participants with TPS ≥1% was defined as the time from randomization to either the date of disease recurrence or death (whatever the cause) as assessed by the investigator. Recurrence of disease was defined as local regional recurrence, a distant (metastatic) recurrence, or a second primary cancer. Occurrence of a second extra-pulmonary malignancy was considered to be an event.
Time Frame: Up to approximately 84 months
Population: All randomized PDL-1 strong positive participants with TPS ≥1%. One participant randomized to the study in error did not provide informed consent and was not included. No data was collected on this participant.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 357 | 355
Months | 58.7 [46.2 to 76.7] | 42.8 [35.0 to 57.8]
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Other; p = 0.01327, Regression, Cox; One-sided p-value was based on the permutation test with multivariate Cox regression model; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 0.97] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death.
Time Frame: Up to approximately 132 months
Reporting Status: Not Posted, anticipated posting 2028-02

5. Secondary Outcome: OS in PDL-1 Strong Positive Participants With TPS ≥50%
Description: OS in PDL-1 Strong Positive Participants with TPS ≥50% was defined as the time from randomization to the date of death.
Time Frame: Up to approximately 132 months
Reporting Status: Not Posted, anticipated posting 2028-02

6. Secondary Outcome: OS in PDL-1 Strong Positive Participants With TPS ≥1%
Description: OS in PDL-1 Strong Positive Participants with TPS ≥1% was defined as the time from randomization to the date of death.
Time Frame: Up to approximately 132 months
Reporting Status: Not Posted, anticipated posting 2028-02

7. Secondary Outcome: Lung Cancer Specific Survival (LCSS)
Description: LCSS was defined as the time from randomization to the date of death (due to lung cancer specifically).
Time Frame: Up to approximately 132 months
Reporting Status: Not Posted, anticipated posting 2028-02

8. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 22 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 580 | 581
Participants | 556 | 529

9. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 580 | 581
Participants | 116 | 34

10. Other Pre Specified Outcome: DFS at 68 Months
Description: as for outcome 1
Time Frame: Up to approximately 68 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 590 | 587
Months | 53.6 [39.2 to NA] — NA = Upper limit DFS was not reached at the time of last disease assessment due to insufficient number of participants with events. | 42.0 [31.3 to NA] — NA = Upper limit DFS was not reached at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Other; p = 0.00143, Regression, Cox; One-sided p-value was based on the permutation test with multivariate Cox regression model; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.63 to 0.91] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 86 months
Description: All-cause mortality was reported on all randomized participants. Serious and non-serious adverse events were reported on all randomized participants who received at least one dose of study treatment. One participant randomized to the study in error did not provide informed consent and was not included. No data was collected on this participant.
Arm/Group | Pembrolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 136/590 | 154/587
Serious Adverse Events (participants affected / at risk) | 142/580 | 90/581
Other Adverse Events (participants affected / at risk) | 510/580 | 458/581
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=580) | Placebo (N=581)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (3) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 5 (7) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (3) | 0 (0)
Hypophysitis (Endocrine disorders) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (3) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (5) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 7 (11) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Asthenia (General disorders) | 2 (2) | 1 (1)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 3 (3)
Sudden death (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (3) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (4) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 13 (15) | 9 (11)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (2)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision site discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0)
Troponin T increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Retrograde amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (3)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (2)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=580) | Placebo (N=581)
Hyperthyroidism (Endocrine disorders) | 62 (65) | 17 (18)
Hypothyroidism (Endocrine disorders) | 120 (148) | 27 (29)
Constipation (Gastrointestinal disorders) | 35 (38) | 41 (53)
Diarrhoea (Gastrointestinal disorders) | 104 (179) | 82 (160)
Nausea (Gastrointestinal disorders) | 52 (64) | 37 (48)
Asthenia (General disorders) | 44 (66) | 32 (39)
Fatigue (General disorders) | 96 (131) | 89 (118)
Influenza like illness (General disorders) | 34 (39) | 32 (36)
Pyrexia (General disorders) | 31 (34) | 32 (48)
Nasopharyngitis (Infections and infestations) | 50 (65) | 32 (44)
Upper respiratory tract infection (Infections and infestations) | 52 (63) | 55 (68)
Alanine aminotransferase increased (Investigations) | 46 (75) | 34 (42)
Aspartate aminotransferase increased (Investigations) | 41 (61) | 31 (40)
Blood creatinine increased (Investigations) | 38 (60) | 32 (52)
Weight decreased (Investigations) | 39 (59) | 25 (36)
Weight increased (Investigations) | 132 (260) | 168 (314)
Decreased appetite (Metabolism and nutrition disorders) | 41 (49) | 26 (28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 107 (152) | 72 (99)
Back pain (Musculoskeletal and connective tissue disorders) | 45 (51) | 46 (57)
Myalgia (Musculoskeletal and connective tissue disorders) | 37 (47) | 15 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 31 (38)
Headache (Nervous system disorders) | 45 (67) | 46 (60)
Paraesthesia (Nervous system disorders) | 18 (19) | 32 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 87 (101) | 98 (130)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 66 (87) | 72 (91)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 32 (52) | 15 (20)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 37 (46) | 15 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 31 (34) | 21 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 125 (167) | 74 (115)
Rash (Skin and subcutaneous tissue disorders) | 49 (69) | 29 (37)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 43 (62) | 20 (27)
Hypertension (Vascular disorders) | 67 (160) | 74 (184)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 30 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT02504372/Prot_SAP_000.pdf